CLINICAL TRIAL: NCT06882928
Title: Applications of Ultrasound and Physical Parameters in Assessing Fall Risk Among Patients With Knee Osteoarthritis: A Prospective Cohort Study
Brief Title: Applications of Ultrasound and Physical Parameters in Assessing Fall Risk in Patients With Knee Osteoarthritis
Acronym: UPPFR-KneeOA
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Clinical Trial Center (Other)
Responsible Party: Sponsor-Investigator, National Taiwan University Clinical Trial Center, physical therapist, National Taiwan University Hospital
Organization: National Taiwan University Hospital (Other)
Other Study IDs: 202501047RINA
Record Dates: First submitted 2025-02-25; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis; Ultrasound Exams; Fall Risk; Sarcopenia in Elderly
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- knee osteoarthritis: Males and females aged 60 and above must have a clinically confirmed diagnosis of knee osteoarthritis.

SUMMARY:
Falls are a significant issue for patients with knee osteoarthritis, as they can lead to hospitalization or even more severe consequences. Therefore, it is crucial to assess fall risk early in rehabilitation clinics. Sarcopenia, which is the reduction of muscle mass, increases the risk of falls. This study involved 250 adults with knee osteoarthritis, using a technology called POCUS to assess muscle mass, combined with other tests to track fall incidents over three months. The study is expected to find correlations between falls and factors like muscle mass and grip strength. This information can help doctors better predict which patients are at risk of falling and take preventive measures early. Future research will explore the effectiveness of different prevention strategies.

DETAILED DESCRIPTION:
Background

Falls represent a significant health issue for patients with knee osteoarthritis, potentially leading to hospitalization, disability, or even death. Early screening for fall risk in rehabilitation clinics is crucial; however, challenges arise due to time constraints and individual differences among patients. Sarcopenia, characterized by a reduction in muscle mass, is closely associated with an increased risk of falls, and point-of-care ultrasound (POCUS) offers a non-invasive and effective tool for assessing muscle mass.

Methods

This prospective study involved 250 adults with knee osteoarthritis attending the orthopedic physical therapy outpatient department at National Taiwan University Hospital. POCUS technology was utilized to evaluate muscle mass, complemented by grip strength tests, lower limb strength assessments, self-reported fall risk questionnaires, sarcopenia assessments, get-up-and-go tests, thirty-second sit-to-stand tests, general nutrition screening for malnutrition, and bioimpedance analysis. A three-month follow-up study was conducted to monitor fall incidents.

Expected Results

During the three-month follow-up, it is anticipated that a certain proportion of participants will experience fall incidents. Significant correlations are expected to be identified between fall incidents and various measurements, including muscle mass assessed by POCUS, grip strength, lower limb strength, self-reported fall risk scores, sarcopenia assessments, get-up-and-go tests, thirty-second sit-to-stand tests, the geriatric nutritional risk index, and bioimpedance analysis. Differences between the fall group and the non-fall group on these variables will also be statistically significant, indicating that the combination of POCUS technology and other clinical assessment indicators enhances the predictive ability regarding fall risk in patients with knee osteoarthritis.

Future Clinical Applications

The integration of POCUS technology with other clinical assessment indicators may be applied in rehabilitation outpatient settings to screen for fall risk in adults with knee osteoarthritis, facilitating early intervention and prevention. Future research will investigate the effectiveness of various intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 60 and above, who are willing to sign an informed consent form.
2. Participants must have a clinically confirmed diagnosis of knee osteoarthritis.
3. Participants must have received at least one treatment in the outpatient rehabilitation department during the study period.
4. Participants must be able to walk independently, even with the aid of assistive devices.

Exclusion Criteria:

1. Individuals who have undergone lower limb surgery or have significant lower limb deformities.
2. Individuals with severe cognitive impairment who are unable to understand or comply with the study procedures.
3. Individuals who cannot communicate in a language understandable by the research team.
4. Individuals with severe comorbidities that affect assessment or treatment (e.g., unable to safely complete assessments or treatments).
5. Individuals planning to undergo knee surgery during the study period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants eligible for the study include males and females aged 60 and above who are willing to sign an informed consent form, have a clinically confirmed diagnosis of knee osteoarthritis, have received at least one treatment in the outpatient rehabilitation department during the study period, and can walk independently, even with the use of assistive devices.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-03-24 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fall Incident Tracking | Three-month period
  Participants will be monitored for fall incidents over a three-month period, and the accuracy of the model predictions will be analyzed.

SECONDARY OUTCOMES:
Grip strength testing | Baseline grip strength
  Measures the maximum strength of hand and forearm muscles using a hand dynamometer. It reflects overall muscle function and the ability to perform daily tasks. Results are reported in kilograms or pounds.
POCUS Assessment | Baseline POCUS Assessment
  Point-of-care ultrasound is used to measure participants' muscle mass
Sarcopenia Risk Assessment Questionnaire (SARC-F) | Baseline Sarcopenia Risk Assessment Questionnaire (SARC-F)
  An assessment tool designed to determine the risk of sarcopenia in individuals. Scale: The SARC-F consists of five questions scored from 0 to 10, with higher scores indicating a greater risk of sarcopenia.
Bioelectrical Impedance Analysis (BIA) Measurement | Baseline BIA measurement
  Conduct bioelectrical impedance measurements to assess body composition, including fat mass and lean body mass.
  Unit of Measure: Results are typically presented in kilograms and percentage for fat mass and lean body mass.
Knee extension strength testing | Baseline knee extension strength testing
  Assesses the strength of the quadriceps by measuring the force exerted during knee extension against resistance, helping evaluate functional mobility. Results can be quantified as force or estimated one-repetition maximum.
Timed Up and Go (TUG) Test | Baseline Timed Up and Go (TUG) Test
  Evaluates mobility and balance by timing how long it takes a participant to rise from a chair, walk three meters, turn, and sit down. Longer times suggest a higher fall risk, especially in older adults.
30-Second Sit-to-Stand Test | Baseline 30-Second Sit-to-Stand Test
  Counts how many times a participant can stand from sitting in 30 seconds. It assesses lower body strength and endurance, with higher counts indicating better functional ability.
Falls Efficacy Scale-International (FES-I) | Baseline Falls Efficacy Scale-International (FES-I)
  A scale that measures the concern about falling during daily activities. Scale: The FES-I includes 16 items scored from 16 to 64, where higher scores indicate greater concern about falling.
Body weight measurement | Baseline body weight measurement
  Measure the body weight of participants using a calibrated scale. Unit of Measure: Kilograms or pounds.
Height Measurement | Baseline height measurement
  Record the participant's height using a stadiometer. Unit of Measure: Meters or centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes